CLINICAL TRIAL: NCT06147323
Title: University of Roehampton
Brief Title: Impact of High Fiber and Vegetal Protein Diet on Gut Health and Immunity Biomarkers in Prediabetic Patients
Acronym: PreVegDiet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Collaborators: Universitat Autonoma de Barcelona (Other); University College Cork (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, Associate Professor in Nutrition and Health, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LSC 23/388
Record Dates: First submitted 2023-11-14; First posted 2023-11-27 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Healthy Diet group (Active Comparator): Participants aged 18-65 years in general good health will be following the Eatwell booklet advice*and NICE/NHS guidelines (https://www.nice.org.uk/).
  Interventions: Other: Normal Healthy Diet
- Placebo Group (Placebo Comparator): Participants aged 18-65 prediabetics will take 2 capsules/day (750mg Maltodextrin placebo comparator) before each of the two main meals without any advice on the diet to follow.
  Interventions: Other: Placebo Diet Group
- Seaweed Group (Active Comparator): Participants aged 18-65 prediabetics will take 2 seaweeds brown extract capsules/day (information detailed in the safety product sheet, total dose of 700 mg before each of the two main meals. All participants will be advised on product storage and use conditions prior to use to ensure product consistency throughout the period of the study.
  Interventions: Dietary Supplement: Seaweed Group

INTERVENTIONS:
Other: Normal Healthy Diet — Participants aged 18-65 years in general good health will be following the Eatwell booklet advice*and NICE/NHS guidelines (https://www.nice.org.uk/).
  Other Names: Eatwell diet Control
  Arms: Normal Healthy Diet group
Dietary Supplement: Seaweed Group — Participants aged 18-65 prediabetics will take 2 seaweeds brown extract capsules/day (information detailed in the safety product sheet, total dose of 700 mg before each of the two main meals. All participants will be advised on product storage and use conditions prior to use to ensure product consistency throughout the period of the study.
  Arms: Seaweed Group
Other: Placebo Diet Group — Participants aged 18-65 prediabetics will take 2 capsules/day (750mg Maltodextrin placebo comparator) before each of the two main meals without any advice on the diet to follow.
  Arms: Placebo Group

SUMMARY:
The research area that focuses on the links between nutrition and health, nutrition and the immune system as well as nutrition-related public health interventions, which often falls into the gap between the agricultural and health domains. The rationale of this project is to study the influence of beneficial diets on the immune system of pre-diabetic patients and its potential to counteract infections. A clinical, an in vitro (cell systems) and an in vivo (animal model) approach will be used to study the influence of a seaweed bioactive supplement and a diet rich in components from a Mediterranean diet on a Salmonella typhimurium infection in prediabetic subjects. At the end of this project, we will provide evidence on the potential of these nutritional interventions to counteract infection, which are of high relevance to the society to reduce the burden of type 2 diabetes (T2DM) and obesity. This research is part of an ongoing research project funded by the Research State Agency (Spain), Health Research Board (HRB, Ireland) and the Medical Research Council (MRC-UKRI, UK) via the NUTRIMMUNE' Grant of the Joint Programming Initiative a Healthy Diet for a Healthy Life (JPI-HDHL).

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effects of different diets on gut health, immune and metabolic markers, in individuals aged between 18-65 years who are defined as pre-diabetics and adults in general good health.

About 45 volunteers will take part in this study and they will then be randomly assigned a volunteer number and placed in one of three study group for a total of 12 weeks:

1. Normal Healthy Diet group (N=15): Participants aged 18-65 years in general good health will be following the Eatwell booklet advice*and NICE/NHS guidelines (https://www.nice.org.uk/).
2. Placebo group (N=15): Participants aged 18-65 prediabetics will take 2 capsules/day (750mg Maltodextrin placebo comparator) before each of the two main meals without any advice on the diet to follow.
3. Seaweed Group.: Participants aged 18-65 prediabetics will take 2 seaweeds brown extract capsules/day (information detailed in the safety product sheet, total dose of 700 mg before each of the two main meals. All participants will be advised on product storage and use conditions prior to use to ensure product consistency throughout the period of the study.

At baseline (week 0), week 6, week 12 and week 16, volunteers will be required to visit the University of Roehampton to provide fasted blood, saliva, stool and first pass urine samples and have blood pressure, body fat and weight measured.

During the study period, they will be asked to complete some questionnaire to assess your gastrointestinal symptoms along with daily stool habits and diet habits.

ELIGIBILITY:
Inclusion criteria

* Adults aged between 18 and 60 years, with
* Fasting blood glucose level of 5.6-6.9mmol/L or impaired HbA1c (HbA1c level of 5.7%-6.4%)
* Fasting blood glucose level below 5.6mmol/L or HbA1c level below 5.7%.
* For intervention purposes, eligible participants are also required to have a mobile phone and be able to read and speak English.

Exclusion criteria

* People with a current diagnosis or clinical history of T2DM
* People with comorbid conditions that may limit participation in the study, such as a history of an acute cardiovascular event, uncontrolled hypertension, cancer or major psychiatric or cognitive problems.
* People who are already participating in a weight loss programme
* People receiving drug treatment for pre-diabetes (eg, metformin)
* People with a history of long-term use of medicines known to influence glucose metabolism (eg, corticosteroids)
* People with elevated liver enzymes (alanine aminotransferase ≥300 IU/L, aspartate aminotransferase ≥300 IU/L)
* People who take antibiotics or bacterial agents (Probiotics) within 1 month
* Pregnant women, women ready for pregnancy, and nursing mothers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2026-08-12 (Estimated)

PRIMARY OUTCOMES:
Changes in blood glucose levels | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effects of dietary intervention on blood glucose levels of pre-diabetics
Changes in insulin sensitivity | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effects of dietary intervention on insulin levels of pre-diabetics
Changes in gut microbiome | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effects of dietary intervention on gut microbiome of pre-diabetics
Changes in pro and anti-inflammatory biomarkers | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effects of dietary intervention on immunity of pre-diabetics
Changes in metabolic profile | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effects of dietary intervention on metabolic signature of pre-diabetics
Changes in dietary habits | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effects of dietary intervention on dietary habits of pre-diabetics
Changes in blood pressure | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effects of dietary intervention on blood pressure of pre-diabetics
Changes in quality of life | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effects of dietary intervention on quality of life of pre-diabetics

CONTACTS AND LOCATIONS:
Overall Officials: ADELE COSTABILE, Dr, Study Director — University of Roehampton
Locations (1):
- Health Sciences Research Centre, Life Sciences Department, University of Roehampton, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Studies website — https://discover-the-secret-of-good-health.weebly.com